CLINICAL TRIAL: NCT01405326
Title: The Effect of Six Months Adalimumab Treatment on Sick Leaves and Retirement in Patients With Rheumatoid Arthritis Who Are at a Risk of Losing Their Ability to Work
Brief Title: REstore Working Ability in RheumatoiD Arthritis
Acronym: REWARD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Rheumatological Center of Helsinki (Network)
Collaborators: Abbott (Industry)
Responsible Party: Kari Eklund MD, Chief of medical affairs, The Rheumatological Center of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: RE100002011
Record Dates: First submitted 2011-06-30; First posted 2011-07-29 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; biological therapy; adalimumab; ability to work; sick leaves
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab (Experimental): Adalimumab treatment for 6 months
  Interventions: Biological: adalimumab
- Pacebo (Placebo Comparator): Corresponding placebo for active treatment group
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — 40mg sc. every two weeks for six months
  Other Names: Humira

SUMMARY:
The purpose of the study is to assess whether a 6-month treatment with adalimumab added on the treatment with conventional antirheumatic drugs (DMARD) will decrease the number of days on sick leave compared to placebo. In addition, the cost-effectiveness and cost-utility of the intervention compared to the conventional treatment is evaluated, and the patients who benefit most are characterized.

DETAILED DESCRIPTION:
In spite of the improved medical treatment, rheumatoid arthritis (RA) is still causing both significant morbidity and marked loss of work productivity. Short periods of work inability, i.e., sick leaves represent a significant part of the socioeconomic burden of RA. The study is a randomized, controlled double blind multi-center study. 160 patients of 25 to 55 years of age with recent-onset (≤2 years from diagnosis) RA who have been treated with a combination of conventional antirheumatic drugs but have an inadequate response to treatment and are at the risk of losing their ability to work, are enrolled. The patients should be biologic-naïve. Their RA should be active, but not so active that the conventional criteria for biologic therapy would be fulfilled. The subjects are randomized at 1:1 ratio to receive either adalimumab (40 mg every two weeks) or placebo for 6 months added on their concurrent antirheumatic therapy. The RA-related sickness absence and clinical response will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of RA according to the 1987 revised American College of Rheumatology (ACR) criteria
2. Time from diagnosis of RA < 2 years
3. Age 25-55 years
4. Active RA with at least 3 active joints (tender and/or swollen joints)
5. Stable DMARD combination treatment for more than 3 months
6. At least one of the following

   * Rheumatoid factor positive
   * One or more erosions in x-rays of the hands and feet
   * Anti-citrulline antibodies positive
7. At least other of the following

   * HAQ-index 0.5 or more
   * Patient or physician evaluation of RA activity >25 mm (VAS 0-10 cm)
8. Patient has been steadily in work-life for at least one year and is currently working or on sick- leave but not applying for pension
9. Patient feels that he/she will likely have to be off-work during the following 6 months due to his/her RA
10. Patient must be willing and able to provide written informed consent for the trial
11. Each female subject must agree to use a medically accepted method of contraception while receiving study medication

Exclusion Criteria:

1. A subject must not have a history of biological drug use for RA
2. A subject must not have evidence of active or latent tuberculosis,
3. A subject must not have any history of lymphoproliferative disease or malignancy within the previous 5 years
4. A subject must not have any other condition, that according to the investigator's judgment makes him or her non-eligible for anti-TNF use
5. A subject must not have any inflammatory rheumatic disease other than RA
6. A subject must not have received any other investigational agents within 30 days prior to baseline visit, and must not receive them during the current trial
7. A female subject must not be pregnant or breast-feeding or planning pregnancy during the study
8. A subject must not have had a major surgery within one month prior to study entry and must not have a scheduled operation during the 6-month follow up
9. A subject must not have any clinically significant condition or situation, other than the condition being studied, that in the opinion of the investigator would interfere with the optimal participation in the trial.
10. A subject must not fulfill the criteria for reimbursement for biologics for RA and he/she would not normally be prescribed a biological drug according to physicians discretion and national treatment guidelines
11. A patient must not be currently on reimbursed rehabilitation period, or such period must not be scheduled for the next six months

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Number of lost work days due to RA during the 6-month follow up. | 6 months

SECONDARY OUTCOMES:
Change in health-related quality of life as measured by the EQ-5D index over the 6-month follow up | baseline and 6 months
Change in functionality assessed by the HAQ over the 6-month follow up | baseline and 6 months
Change in disease activity measured with DAS28 with CRP and ESR over the 6-month follow up | baseline and 6 months
Work Productivity and Activity Impairment Questionnaire (WPAI) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kari K Eklund, MD, Principal Investigator — The Rheumatological Center of Helsinki
Locations (4):
- Finland (4):
  - Helsinki University Central Hopsital, Helsinki
  - Lappland Central Hospital, Rovaniemi
  - Tampere University hospital, Rheumatology Centre, Tampere
  - The Turku Universitry Central Hopsital, Turku